CLINICAL TRIAL: NCT06996119
Title: Pilot Study of Emapalumab With Post-Transplant Cyclophosphamide as Graft-Versus-Host Disease Prophylaxis for Reduced-Intensity Allogeneic Hematopoietic Cell Transplantation
Brief Title: Emapalumab With Post-Transplant Cyclophosphamide, Tacrolimus and Mycophenolate Mofetil for the Prevention of Graft-versus-Host Disease After Donor Reduced-Intensity Hematopoietic Cell Transplant
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23822; NCI-2025-03603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23822 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Graft Versus Host Disease; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Graft vs Host Disease; Myelodysplastic Syndromes | interventions — Specimen Handling; Busulfan; Cyclophosphamide; Emapalumab; fludarabine; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Melphalan; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (emapalumab, cyclophosphamide) (Experimental): Patients receive fludarabine IV on days -7 to -3 and melphalan IV over 1 hour on day -2 or busulfan IV on days -7 and -6 and fludarabine IV on days -7 to -2. Patients receive HCT infusion on day 0 per institutional standards of practice. Patients also receive emapalumab IV over 1 hour on days -8. -1, -7, 14 and 21, cyclophosphamide IV on days 3 and 4, tacrolimus IV or PO on days 5-95, mycophenolate mofetil IV or PO on days 5-35. Additionally, patients undergo chest CT and ECHO or MUGA at baseline and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Busulfan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Biological: Emapalumab; Drug: Fludarabine; Procedure: Hematopoietic Cell Transplantation; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Drug: Mycophenolate Mofetil; Other: Questionnaire Administration; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Procedure: Computed Tomography — Undergo chest CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Emapalumab — Given IV
  Other Names: Anti-IFN gamma Monoclonal Antibody NI-0501; Anti-IFNg mAb NI-0501; Anti-interferon gamma Monoclonal Antibody NI-0501; Emapalumab-lzsg; Gamifant; NI 0501; NI-0501; NI0501
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Hematopoietic Cell Transplantation — Given infusion
  Other Names: HCT; Hematopoietic Stem Cell Infusion; HEMATOPOIETIC STEM CELL TRANSPLANT; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; Stem Cell Transplantation, NOS
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: CellCept; MMF
Other: Questionnaire Administration — Ancillary studies
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius

SUMMARY:
This phase I trial tests the safety, side effects and effectiveness of emapalumab with post-transplant cyclophosphamide, tacrolimus, and mycophenolate mofetil in preventing graft-versus-host disease (GVHD) in patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) after reduced-intensity donor (allogeneic) hematopoietic cell transplant (HCT). Giving chemotherapy, such as fludarabine, melphalan, or busulfan, before a donor [peripheral blood stem cell] transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When healthy stem cells for a donor are infused into a patient (allogeneic HCT), they may help the patient's bone marrow make more healthy cells and platelets. Allogeneic HCT is an established treatment, however, GVHD continues to be a major problem of allogeneic HCT that can complicate therapy. GVHD is a disease caused when cells from a donated stem cell graft attack the normal tissue of the transplant patient. Emapalumab binds to an immune system protein called interferon gamma. This may help lower the body's immune response and reduce inflammation. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid and may kill cancer cells. It may also lower the body's immune response. Tacrolimus is a drug used to help reduce the risk of rejection by the body of organ and bone marrow transplants. Mycophenolate mofetil is a drug used to prevent GVHD after organ transplants. It is also being studied in the prevention of GVHD after stem cell transplants for cancer, and in the treatment of some autoimmune disorders. Mycophenolate mofetil is a type of immunosuppressive agent. Giving emapalumab with post-transplant cyclophosphamide, tacrolimus and mycophenolate mofetil may be safe, tolerable and/or effective in preventing GVHD in patients with AML or MDS after a reduced-intensity allogeneic HCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and describe the toxicity profile of adding emapalumab to post-transplant cyclophosphamide (PTCy)-based graft-versus-host disease (GVHD) prophylaxis by day 28 post reduced-intensity hematopoietic cell transplantation (HCT).

SECONDARY OBJECTIVES:

I. Estimate activity of emapalumab, PTCy, tacrolimus (tacro) and mycophenolate mofetil (MMF) acute GVHD (aGVHD) prophylaxis, by cumulative incidence of aGVHD (grade 2-4) at day +100.

II. Estimate cumulative incidence of chronic GVHD (cGVHD) at 1-year post-HCT. III. Estimate overall survival (OS) and progression-free survival (PFS) at 1- year post-transplant.

IV. Estimate GVHD-free relapse-free survival (GRFS) at 1-year post-HCT. V. Estimate cumulative incidence of relapse/disease progression, and non-relapse mortality (NRM) at day +100 and 1-year post-HCT.

VI. Estimate the rate of grade 2 or higher infection at 100 days. VII. Assess time to engraftment (platelets and neutrophils).

EXPLORATORY OBJECTIVES:

I. Evaluate free emapalumab levels by serial blood sampling and assess association with severe aGVHD incidence.

II. Determine levels of interferon gamma (IFNgamma)-related inflammatory cytokines (CXCL-9 and CXCL-10) by serial sampling and assess association with free emapalumab levels and incidence of grade 3-4 aGVHD.

III. aGVHD biomarkers per Mount Sinai Acute GVHD International Consortium (MAGIC) criteria on days + 1, +7, +14 and +28.

IV. Describe the kinetics of immune cell recovery (B, T, natural killer [NK] cells) at days 30, +100, +180 and +365 post-HCT in peripheral blood.

V. Evaluate patient quality of life at baseline then on day +100, 6 months, and 1-year post-HCT using patient reported outcomes of Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT).

VI. Obtain a preliminary estimate of gut microbiome diversity at baseline (preferably before fludarabine administration), and then on days +14, +28, +60, and +100 after HCT.

OUTLINE:

Patients receive fludarabine intravenously (IV) on days -7 to -3 and melphalan IV over 1 hour on day -2 or busulfan IV on days -7 and -6 and fludarabine IV on days -7 to -2. Patients receive HCT infusion on day 0 per institutional standards of practice. Patients also receive emapalumab IV over 1 hour on days -8. -1, -7, 14 and 21, cyclophosphamide IV on days 3 and 4, tacrolimus IV or orally (PO) on days 5-95, mycophenolate mofetil IV or PO on days 5-35. Additionally, patients undergo chest computed tomography (CT) and echocardiography (ECHO) or multigated acquisition scan (MUGA) at baseline and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 100 days after HCT, then at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 18 years and ≤ 75 years

  * Note: Patients > 70 years of age must have Karnofsky performance status ≥ 80% and HCT-comorbidity index (CI) ≤ 2
* Karnofsky performance status ≥ 70%
* Patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) in complete remission with bone marrow (BM) blast of < 5%. AML must be negative for minimal residual disease (MRD-)
* Planned to undergo reduced-intensity conditioning (RIC) with either fludarabine/melphalan (Flu/Mel) or busulfan/fludarabine (Bu/Flu) regimens prior to an allogeneic HCT using a mobilized peripheral blood stem cell (PBMC) graft from an 8/8 match related/unrelated donor (A, B, C, DR by high resolution typing)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN
* Creatinine clearance of ≥ 60 mL/min per 24-hour urine test or the Cockcroft-Gault formula
* Left ventricular ejection fraction (LVEF) ≥ 50%

  * Note: To be performed within 30 days prior to day 1 of protocol therapy
* Bazett's correction formula (QTcB) ≤ 480 ms
* If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) (diffusion capacity) ≥ 50% of predicted (corrected for hemoglobin).
* If unable to perform pulmonary function tests: Oxygen (O2) saturation > 92% on room air
* Seronegative for HIV antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) OR

  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* QuantiFERON-TB Gold+

  * Administer tuberculosis prophylaxis to patients at risk for tuberculosis, or known to have a positive purified protein derivative (PPD) test result, or positive interferon gamma (IFNγ) release assay
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 180 days post-HCT

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior allogeneic HCT
* Other cancer therapies (chemotherapy, radiation, biologics) are not allowed within two weeks of starting HCT conditioning; however targeted agents for underlying hematologic malignancies may be continued up to one day before conditioning, including, but not limited to:

  * FLT3 inhibitors
  * IDH1/2 inhibitors
  * Menin inhibitors
  * ABL-BCR inhibitors
  * BCL-2 inhibitors
  * Hydroxyurea
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Psychological issues, no appropriate caregivers identified, or non-compliant to medication
* Clinically significant uncontrolled illness
* Active uncontrolled infections (bacterial, viral, fungal). Infections are considered controlled if appropriate therapy has been initiated and, at the time of screening, no signs of infection are present
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-05-25 (Estimated); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher adverse events (AEs) | From starting the first emapalumab dose to the first observation of a primary safety endpoint (PSE) event or day 28 post-hematopoietic cell transplantation (HCT), whichever comes first
  Will be based on Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0, with the exception of infections which ill be graded based on the Report of the Bone Marrow Transplant (BMT) Clinical Trials Network (CTN) Infections Disease Technical Committee. The toxicity/AE information recorded on each subject will include type, severity, duration, and attribution/ association with the study regimen. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection.
Incidence of severe infusion reaction | From starting the first emapalumab dose to the first observation of a PSE event or day 28 post-HCT, whichever comes first
  Will be defined as grade 4 per CTCAE v 5.0 after receiving the first or second dose of emapalumab. The toxicity/AE information recorded on each subject will include type, severity, duration, and attribution/ association with the study regimen. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection.
Incidence of primary graft failure | From starting the first emapalumab dose to the first observation of a PSE event or day 28 post-HCT, whichever comes first
  Will be defined as the failure to achieve an absolute neutrophil count of 500/ul or more for 3 days and donor chimerism of less than 5%. Will be calculated using the competing risk method as described by Gooley et al. (1999).
Non-relapse mortality (NRM) | From starting the first emapalumab dose to the first observation of a PSE event or day 28 post-HCT, whichever comes first
  Will be calculated using the competing risk method as described by Gooley et al. (1999).

SECONDARY OUTCOMES:
Incidence of grade 2-4 acute graft-versus-host-disease (aGVHD) | At day 100
  Will be calculated using the competing risk method as described by Gooley et al. (1999).
Incidence of grade 3 or higher AEs | From day 29 to day 100
  Will be defined by CTCAE v 5.0 with the exception of infections which will be graded based on the Report of the BMT CTN Infectious Disease Technical Committee. The toxicity/AE information recorded on each subject will include type, severity, duration, and attribution/ association with the study regimen. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection.
Overall survival | From the day of stem cell infusion until death, assessed up to 1 year
  Will be calculated using the Kaplan-Meier method.
Progression free survival | From the date of stem cell infusion to the date of death, disease relapse/progression, whichever occurs first, assessed up to 1 year
  Will be calculated using the Kaplan-Meier method.
GVHD relapse-free survival (GRFS) | From the start of HCT to grade III-IV aGVHD, chronic GVHD, requiring systemic treatment, relapse, or death from any cause, whichever occurs first, assessed up to 1 year
  Will be calculated using the Kaplan-Meier method.
Relapse/progression | From day of stem cell infusion (day 0) and at 100 days and at 1 year
  Will be calculated using the Kaplan-Meier method.
NRM | From date of stem cell infusion until non-disease related death, assessed up to 1 year
  Will be defined as death occurring in a patient from causes other than relapse or progression. The toxicity/AE information recorded on each subject will include type, severity, duration, and attribution/ association with the study regimen. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection.
Incidence of aGVHD | From day 0 (date of stem cell infusion) through 180 days post-transplant
  Will be calculated using the competing risk method as described by Gooley et al. (1999).
Incidence of chronic GVHD | From day 80 through 1 year post-transplant
  Will be evaluated and scored according to National Institutes of Health Consensus Staging. Will be calculated using the competing risk method as described by Gooley et al. (1999).
Incidence of infection | From day -7 to day 100 post-transplant
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any, according to the Report of the BMT CTN Infectious Disease Technical Committee. The toxicity/AE information recorded on each subject will include type, severity, duration, and attribution/ association with the study regimen. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection.
Absolute neutrophil count recovery | Up to 1 year
  Will be defined as neutrophils >= 0.5 x 10^3/uL achieved and sustained for 3 consecutive lab values on different days with no subsequent decline.
Platelet recovery | Up to 1 year
  Will be defined as platelets >= 20 K/uL independent of platelet transfusion support (date should reflect no transfusions in previous 7 days, and the first of 3 consecutive lab values on different days).

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States